CLINICAL TRIAL: NCT03935139
Title: Monitoring of the Bone Free Flaps With Microdialysis
Acronym: MTM2018
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0023
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Flap Necrosis
Keywords: microdialysis; bone free flap; fibula; iliac crest
MeSH Terms: interventions — Glycerol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: glucose measurement — Glucose values will be recorded during 5 days as following : every hour at day 0, every 2 hours at day 1, every 3 hours at days 2 to 5.
Biological: lactacte measurement — Lactate values will be recorded during 5 days as following : every hour at day 0, every 2 hours at day 1, every 3 hours at days 2 to 5.
Biological: pyruvate measurement — pyruvate values will be recorded during 5 days as following : every hour at day 0, every 2 hours at day 1, every 3 hours at days 2 to 5.
Biological: glycerol measurement — glycerol values will be recorded during 5 days as following : every hour at day 0, every 2 hours at day 1, every 3 hours at days 2 to 5.
Procedure: Bone free flap monitoring — Bone free flaps will be monitored with a microdialysis catheter directly positioned in bone tissue.

SUMMARY:
Microdialysis is admitted to be reliable by numerous surgeons to monitor flaps. Nevertheless, a few authors reported follow up with microdialysis in bone free flaps, and they all describe the position of the catheter in the surrounding soft tissue muscle which is not the accurate reflect of bone vascularisation. The aim of this study is to determine the lactate/pyruvate ratio mean value in bone free flaps with a microdialysis catheter directly positioned in the bone tissue.

DETAILED DESCRIPTION:
Failure rate of facial reconstructive surgery with bone free flaps varies between 11 and 25%. In case of buried bone free flaps, the follow up is even more difficult. Monitoring methods, such as the implantable Doppler system, laser Doppler flowmetry and microdialysis have been developped in the last 15 years. Ferguson et al. show a false positive rate of 31% with implantable doppler monitoring of buried flaps.

The purpose of this study is to to determine the lactate/pyruvate ratio mean value in bone free flaps with a microdialysis catheter directly positioned in the bone tissue.

ELIGIBILITY:
Inclusion Criteria:

* adult person
* signed informed consent
* head and neck reconstruction with iliac crest or fibula free flap
* patient covered by national health insurance

Exclusion Criteria:

* minor person
* head and neck reconstruction with other types of free flaps than crest or fibula free flap
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of lactate/pyruvate ratio in patients without free flap ischemia | every hour during the day of surgery
  Change from Baseline of lactate/pyruvate ratio in patients without free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without free flap ischemia | every 2 hours at day 1 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients without free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without free flap ischemia | every 3 hours at days 2, 3 , 4 and 5 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients without free flap ischemia

SECONDARY OUTCOMES:
Change from Baseline of lactate/pyruvate ratio in patients without fibula free flap ischemia | every hour during the day of surgery
  Change from Baseline of lactate/pyruvate ratio in patients without fibula free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without fibula free flap ischemia | every 2 hours at day 1 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients without fibula free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without fibula free flap ischemia | every 3 hours at days 2, 3 , 4 and 5 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients without fibula free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without crest free flap ischemia | every hour during the day of surgery
  Change from Baseline of lactate/pyruvate ratio in patients without crest free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without crest free flap ischemia | every 2 hours at day 1 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients without crest free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients without crest free flap ischemia | every 3 hours at days 2, 3 , 4 and 5 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients without crest free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients with free flap ischemia | every hour during the day of surgery
  Change from Baseline of lactate/pyruvate ratio in patients with free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients with free flap ischemia | every 2 hours at day 1 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients with crest free flap ischemia
Change from Baseline of lactate/pyruvate ratio in patients with free flap ischemia | every 3 hours at days 2, 3 , 4 and 5 after surgery
  Change from Baseline of lactate/pyruvate ratio in patients with crest free flap ischemia
Change from Baseline of metabolites rate in patients with free flap ischemia | every hour during the day of surgery
  Metabolites measurement are glucose, lactate , pyruvate and glycerol rates.
Change from Baseline of metabolites rate in patients with free flap ischemia | every 2 hours at day 1 after surgery
  Metabolites measurement are glucose, lactate , pyruvate and glycerol rates.
Change from Baseline of metabolites rate in patients with free flap ischemia | every 3 hours at days 2, 3 , 4 and 5 after surgery
  Metabolites measurement are glucose, lactate , pyruvate and glycerol rates.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Dakpe, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No